CLINICAL TRIAL: NCT01189318
Title: Effects of Seroquel XR (Quetiapine Fumarate Extended-Release) on Sleep Architecture in Patients With Major Depressive Disorder
Brief Title: Effects of Seroquel XR on Sleep Architecture in Patients With Major Depressive Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443C00042
Record Dates: First submitted 2010-08-17; First posted 2010-08-26 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seroquel XR (Experimental): Patients with MDD receives Seroquel XR.
  Interventions: Drug: Quetiapine Fumarate Extended Release
- healthy control (No Intervention)

INTERVENTIONS:
Drug: Quetiapine Fumarate Extended Release — Day 1 50mg, Day 2 50mg, Day 3 150mg, Day 4~28 50~150mg (increments and deduction of 50mg are allowed)
  Arms: Seroquel XR

SUMMARY:
In this study, patients with major depressive disorder (MDD) who have insomnia symptom are treated with Seroquel XR in an open-label manner for a 4-week period with repeated measurements of insomnia symptoms and sleep parameters using polysomnography.

ELIGIBILITY:
Patient Inclusion Criteria:

* Men and women aged between 20 and 65
* Diagnosis of major depressive disorder as assessed by Structured Clinical Interview for DSM-IV (SCID-IV)
* A score of 1 or greater on any of the sleep items (items 4, 5, 6) from the Hamilton Depression Rating Scale (HDRS)
* Provision of written informed consent

Healthy Control Subject Inclusion Criteria:

* Healthy Men and Women aged between 20 and 65
* Provision of written informed consent

Exclusion Criteria:

* Presence of any major physical or neurological illness (e.g.，head trauma， epilepsy，seizure，stroke，cerebral tumor，multiple sclerosis，cerebrovascular disease, narrow-angle glaucoma, drug hypersensitivity，etc.)
* Diagnosis of any Axis I disorder other than major depressive disorder or presence of symptoms requiring hospitalization
* Drug abuse in past 3 months
* Women who are pregnant，breastfeeding, or planning pregnancy
* Contraindications to drugs used in the study (e.g., allergy, intolerance, etc.)
* Unstable medical illness or severe abnormality in laboratory test at screening assessment
* Increase in blood glucose, lipid, and calcium levels at screening
* Low blood pressure at screening assessment
* Intelligence quotient below 80
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
* Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 3 months prior to enrolment
* Previous enrolment or randomisation of treatment in the present study.
* Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* A patient with Diabetes Mellitus
* An absolute neutrophil count (ANC) of <= 1.5 x 10^9 per liter
* Insomnia from other causes of medical or neurological diseases
* Involvement in the planning and conduct of the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
change from baseline Pittsburgh Quality Index total scores at 4 weeks | baseline and 4 weeks
change from baseline Pittsburgh Quality Index total scores at 2 weeks | baseline and 2 weeks
change from baseline Pittsburgh Quality Index total scores at 4 days | baseline and 4 days

SECONDARY OUTCOMES:
change from baseline in sleep architecture measured using polysomnography at 4 weeks | baseline and at 4 weeks
number of participants with adverse events | 4 weeks
number of participants with adverse events | 2 weeks
number of participants with adverse events | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Inkyoon Lyoo, MD, PhD, MMS, Principal Investigator — Ewha Womans University
Locations (1):
- Ewha Womans University Medical Center, Seoul, South Korea